CLINICAL TRIAL: NCT05333094
Title: Comparison Between the Effectiveness of Different Commercial Bracket Brands, Having Roth Prescription and 0.022" Bracket Slot: A Randomized Clinical Trial
Brief Title: Comparison Between the Effectiveness of Different Commercial Bracket Brands
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Salma Khaled Kamal Yacoub, Principle investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUE.REC(32)/12-2020
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Crowding, Tooth, Class I
Keywords: orthodontic bracket brands; torque prescription; tip prescription; levelling and Alignment; Lateral Cephalometric Radiographs; CBCT; VAS
MeSH Terms: conditions — Crowding | interventions — Orthodontic Brackets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single (Outcomes Assessor) Only the outcome assessors will be blind. The patients name will be sealed from pre and post radiographs and study models. Then two assessors will carry out, blindly and independently, the measurements and analysis of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- American orthodontics brackets (Active Comparator): Roth prescription, 0.022" slot size
  Interventions: Other: Brackets
- FANTA brackets (Active Comparator): Roth prescription, 0.022" slot size
  Interventions: Other: Brackets
- MATT brackets (Active Comparator): Roth prescription, 0.022" slot size
  Interventions: Other: Brackets

INTERVENTIONS:
Other: Brackets — Levelling and alignment for the bonded teeth through following the wire sequence: 0.014 NiTi, 16 NiTi, 0.016×0.022 NiTi and 0.017×0.025 StSt. (Wires from American Orthodontics)
  • After levelling and aligning is completed the patient will be referred for the uptake of post intervention records; a standardized dental photograph and CBCT after 6- 9 months)

SUMMARY:
There's a scarcity in literature concerning the comparison of the effectiveness of brackets in its torque and tip ability, the time takes for leveling and alignment comparing between different orthodontic bracket brands, and its effect on the rate of tooth movement. The purpose of this study is to determine, In orthodontic patients with Class I molar relation and teeth crowding, in which different bracket brands will be compared.

DETAILED DESCRIPTION:
Bracket effectiveness can be measured in a variety of ways, including torque, tip, time required for levelling and alignment, bracket failure, and the patient's visual analogue scale. All are viable options; therefore, we want to complete the orthodontic treatment and determine which brackets fulfilled the built-in bracket prescription and achieved success in terms of aesthetics, better smiles, better patient judgement, and function.

ELIGIBILITY:
Inclusion Criteria:

* Patient with full set of permanent teeth
* Male and female (14-19 years old).
* Positive patients' acceptance for the study
* Patients have no history of previous orthodontic treatment.

Exclusion Criteria:

* Patients with enamel or dentin defect or any teeth anomaly will be eliminated.
* Patients having canine or lateral incisors peg shaped will be excluded from the research. - Medically compromised patients
* Patients unable to give an informed consent
* Patient with periodontal disease
* Patient taking long term medication
* Patients with any parafunctional habits (i.e. Bruxism, tongue thrusting, mouth Breathing)

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Tip | From pre to post levelling and alignment (an average of 6 - 8 months)
  The principle investigator will examine pre and post CBCT radiographs in relation to lines and reference planes (measurements in degrees and mm)
torque | 3 months after reaching 19x25 stainless steel wire (an average of 6 - 8 months)
  The principle investigator will examine pre and post CBCT radiographs in relation to lines and reference planes (measurements in degrees and mm)

SECONDARY OUTCOMES:
Levelling and alignment | upto 6 months from the start of orthodontic treatment.
  The incisal edges of the anterior teeth and the buccal cusps of the posterior teeth are placed on the same horizontal level; and alignment is the lining up of teeth of an arch in order to achieve normal contact point relationships will be assessed by measuring Little's Irregularity Index (LII) using study models taken of the patients (measured in mm)

OTHER OUTCOMES:
Pain of intervention | From pre to post levelling and alignment (an average of 6 - 8 months)
  Each patient will fill a questionnaire regarding his treatment experience in a VAS scoring from 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Yehya A. Mostafa, Professor and Chairman, Study Director — Future University in Egypt
Locations (1):
- Future University In Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All Collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication